CLINICAL TRIAL: NCT06440837
Title: Effectiveness of Stress Self-management Health Education Based on IMB Theory Among Nursing Students, Shanxi Province, China
Brief Title: Effectiveness of Stress Self-management Health Education Based on IMB Theory Among Nursing Students
Acronym: IMB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changzhi Medical College (Other)
Responsible Party: Principal Investigator, Dong Xiujuan, research leader, Changzhi Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ChangzhiMC
Record Dates: First submitted 2024-05-28; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Psychological Stress; Nursing Students
Keywords: health education; IMB model; cluster-randomized controlled study
MeSH Terms: conditions — Stress, Psychological; Health Education

STUDY DESIGN:
Intervention Model Description: The random sequence generation will be implemented at the cluster level rather than the individual level to prevent sample contamination. Dormitories meeting the eligibility criteria will be coded and randomly assigned to either the intervention group or the control group. The random assignment will be executed using computer-generated software on a research randomization website, with a 1:1 allocation ratio.
Who Masked: Investigator, Outcomes Assessor
Masking Description: To ensure allocation concealment, an external party using a "third-party" allocation approach will be employed. This involves using a research assistant to maintain allocation concealment. The list of eligible dormitories will be sent to a second research assistant, who will then carry out the sequence generation described above. Neither the researchers nor other research personnel will be aware of the specific dormitory group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- wait-list (No Intervention): participant in this group will not accept any psychological intervention content during experimental period. After the study, the intervention will be distributed for free.
- IMB stress self-management health education (Experimental): Participants in this arm will receive an online "IMB stress self-management health education" program. The health education intervention program contains eight module topics.
  Interventions: Behavioral: IMB stress self-management health education

INTERVENTIONS:
Behavioral: IMB stress self-management health education — The health education intervention program contains eight module topics: stress-related knowledge, the thinking and mentality under stress, social support, take care of your suffering, manage your difficult emotions, acceptance, embrace a better life, ending. One topic or session is delivered by weeks, each session lasting 30-40 minutes.
  Other Names: "information-motivation-behavioral skills" stress self-management health education
  Arms: IMB stress self-management health education

SUMMARY:
The aim of this cluster randomized controlled study is to test the effectiveness of IMB stress self-management health education on nursing students registered in first semester. The main question aims to answer are: Does IMB stress self-management health education program improving stress in nursing students? Researcher will compare wait-list group without any intervention to experimental group which received IMB stress self-management health education, to see if IMB stress self-management health education works to improving stress among nursing students.

Participants will Attend IMB stress self-management health education program once a week for 8 weeks. In addition, complete questionnaires at pre-intervention, post-intervention, 1-month post-intervention, 3-months post-intervention, 6-months post-intervention.

DETAILED DESCRIPTION:
This study intends to select first-year undergraduate nursing students registered in October 2024 at Changzhi Medical College in Shanxi as the sampling population. A total of 120 eligible individual samples in eligible clusters will be screened according to inclusion and exclusion criteria, and the cluster samples will be randomly assigned to either the wait-list group or the intervention group. Participants in wait-list group will not receive any intervention, while participants in intervention group will receive IMB-based stress self-management health education. The intervention will last for 8 weeks, with one module delivers by weeks. Each module will include a 30-40 minute lecture combined with exercises, discussions, and role-playing activities. Measurements will be taken before the intervention, immediately after the intervention, and at 1 month, 3 months, and 6 months post-intervention. These measurements will include the Stress Knowledge Questionnaire, the Multidimensional Scale of Perceived Social Support, the Self-Compassion Scale, the Resilience Scale, and the stress sub-scale of the Depression Anxiety Stress Scale.

The study data will be analyzed using the intention-to-treat (ITT) method. Continuous data will be described using mean (standard deviation) or median (interquartile range), and categorical data will be described using frequency and percentage. Repeated measures ANOVA will be used to compare differences between the two groups before the intervention, immediately after the intervention, and at 1 month, 3 months, and 6 months post-intervention. Generalized linear models (GMM) will be utilized to determine the effects of IMB-based stress self-management health education on the variables immediately post-intervention, and at 1 month, 3 months, and 6 months post-intervention, while controlling for confounding variables. Sensitivity analysis will be performed and reported. The mean estimates will be set with a 95% confidence interval, and the significance level will be set at P < 0.05.

This study aims to explore new low-cost approaches for current college student mental health education, improve stress self-management abilities and stress levels among nursing students, prevent mental disorders, and promote mental health. To ensure the safety of participants throughout the study, the research team will strictly adhere to ethical standards and undergo review and supervision by the ethics committee. Informed consent will be obtained from participants, and their privacy and personal information will be kept confidential, not disclosed or misused. Regular safety monitoring and risk assessments will be conducted. The research protocol will be strictly followed, and psychological counseling services will be provided to participants.

ELIGIBILITY:
Inclusion Criteria:

1. cluster

   * dormitories located in Changzhi Medical College
   * The residents in the dormitory are all nursing students that registered in fist-semester
2. individual

   * Registered in undergraduate nursing program
   * Registered in the first-semester study
   * Have a mobile device that can access internet
   * Voluntarily participated in this study

Exclusion Criteria:

1. cluster

   * The residents in the dormitory are mixed with students from other majors except nursing.
   * The residents in the dormitory are mixed with nursing students from other grade.
2. individual

   * Diagnosed with mental problems or severe physical problems, e.g., depression, generalized anxiety disorder, or diabetes
   * Previous participation in other stress intervention studies

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-10-10 (Estimated); Primary Completion 2025-06-10 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
stress sub-scale of DASS-21 | baseline, immediately after the intervention, 1 month after the intervention, 3 months after the intervention, 6 months after the intervention.
  The DASS-42 is a 42 item self-report scale is designed to measure the emotional states of depression, anxiety and stress. Each of the 42 questions in DASS is scored on a 4-point scale ranging from 0("Did not apply to me at all") to 3("Applied to me very much, or most of the time"). Scores for Stress is calculated by summing the scores for the 14 items: 1, 6, 8, 11, 12, 14, 18, 22, 27, 29, 32, 33, 35, 39. Total score of the stress subscale ranged from 0 to 42, the level of stress can be categorized five level based on total score actually measured: normal (score from 0 to 14), mild (score from 15 to 18), moderate (score from 19 to 25), Sever (score from 26 to 33), extreme sever (score from 34 above), therefore, higher score indicate higher level of stress.

SECONDARY OUTCOMES:
Stress Knowledge Questionnaire | baseline, immediately after the intervention, 1 month after the intervention, 3 months after the intervention, 6 months after the intervention.
  Stress Knowledge Questionnaire (SKQ) is used to assess people's knowledge of stress. The questionnaire is consisting of 7 questions using true/false options as answer.
Stress Mindset Measure-General | baseline, immediately after the intervention, 1 month after the intervention, 3 months after the intervention, 6 months after the intervention.
  Stress Mindset Measure- General is a self-reported instrument used to measure individual's belief toward stress. It is an 8-item tool to address the extent to which an individual adopts a mindset that the effects of stress are enhancing or debilitating. Each item rated in form of 5-Likert scale, ranging from 0=strongly disagree to 4=strongly agree. The item 1, 3, 5, 7 is negative items while the item 2, 4, 6, 8 is positive item. The total score is obtained by reverse scoring the four negative items and then taking the mean of all 8 items. Higher scores represent the mindset that stress is enhancing.
Multidimensional Scale of Perceived Social Support | baseline, immediately after the intervention, 1 month after the intervention, 3 months after the intervention, 6 months after the intervention.
  Multidimensional Scale of Perceived Social Support (MSPSS) is a self-report measure of social support scale that emphasizes individual subjective understanding and feelings. The questionnaire is a 12-item scale which designed to assess three perceived sources of supports: family (Items 3, 4, 8, and 11), friends (Items 6, 7, 9, and 12) and significant others (Items 1, 2, 5, and 10). Each item is scored from 1 (extremely disagree) to 7 (extremely agree). Three level of support can be categorized by the mean scale score. The mean scale score ranged from 1 to 2.9 could be considered low support; a score of 3 to 5 could be considered moderate support; a score from 5.1 to 7 could be considered high support.
Self-Compassion Scale Short Form | baseline, immediately after the intervention, 1 month after the intervention, 3 months after the intervention, 6 months after the intervention.
  The Chinese version of Self-Compassion Scale consists 12 items on five-point Likert scale (0= 'almost never' to 5= 'almost always') to record how often you behave kindly and caring toward yourself in difficult situations. It could be used to test three dimensions of self-compassion: Common Humanity, Mindfulness, and Self-Kindly. Item 2, 4, 5, 8, 11 are reverse scored item. The total score of the instrument ranged from 12 to 60, higher score indicates higher self-compassion, vice versa. The Chinese version SCS-SF exhibit high reliability and validity.
Connor-Davidson Resilience Scale | baseline, immediately after the intervention, 1 month after the intervention, 3 months after the intervention, 6 months after the intervention.
  The 10-item psychological resilience scale is used to measure the ability to cope with illness, stress, failure, etc. The scale is a 5-point Likert (0= 'almost never' to 4= 'almost most') self-reported questionnaire; The total score of the scale is the sum of the response of each item, ranged from 0 to 40; Higher total score indicates higher resilience capacity.

CONTACTS AND LOCATIONS:
Overall Officials: binti Ahmad Norliza, Dr, Study Director — University Putra Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Result] Connor KM, Davidson JR. Development of a new resilience scale: the Connor-Davidson Resilience Scale (CD-RISC). Depress Anxiety. 2003;18(2):76-82. doi: 10.1002/da.10113. PMID 12964174
- [Result] Crum AJ, Salovey P, Achor S. Rethinking stress: the role of mindsets in determining the stress response. J Pers Soc Psychol. 2013 Apr;104(4):716-33. doi: 10.1037/a0031201. Epub 2013 Feb 25. PMID 23437923
- [Result] Zimet GD, Powell SS, Farley GK, Werkman S, Berkoff KA. Psychometric characteristics of the Multidimensional Scale of Perceived Social Support. J Pers Assess. 1990 Winter;55(3-4):610-7. doi: 10.1080/00223891.1990.9674095. PMID 2280326